CLINICAL TRIAL: NCT01471366
Title: What is the Best Way to Take Fish Oil?
Brief Title: Method of Fish Oil Administration on Patient Compliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi, Oxford (Other)
Collaborators: Walgreens (Industry)
Responsible Party: Principal Investigator, Daniel Riche, Principal Investigator, University of Mississippi, Oxford
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: UMO-0003
Record Dates: First submitted 2011-11-10; First posted 2011-11-16 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Adverse Effects
Keywords: Hyperlipidemias; Dyslipidemias; Fatty Acids, Omega-3; Fish Oils
MeSH Terms: conditions — Hyperlipidemias; Dyslipidemias | interventions — Freezing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Frozen capsule (Active Comparator): Two frozen fish oil capsules (300 mg EPA/DHA per capsule) by mouth three times daily with 8 ounces of water without food or dairy products
  Interventions: Dietary Supplement: Frozen capsule
- Capsule with food (Active Comparator): Two room temperature fish oil capsules (300 mg EPA/DHA per capsule) by mouth three times daily with 8 ounces of water with food but no dairy products
  Interventions: Dietary Supplement: Capsule with food
- Capsule without food (Active Comparator): Two room temperature fish oil capsules (300 mg EPA/DHA per capsule) by mouth three times daily with 8 ounces of water with no food or dairy products
  Interventions: Dietary Supplement: Capsule without food
- Capsule with milk (Active Comparator): Two room temperature fish oil capsules (300 mg EPA/DHA per capsule) by mouth three times daily with 8 ounces of milk with no food or additional dairy products
  Interventions: Dietary Supplement: Capsule with milk

INTERVENTIONS:
Dietary Supplement: Frozen capsule — Two frozen fish oil capsules (300 mg EPA/DHA per capsule) by mouth three times daily with 8 ounces of water without food or dairy products.
  Other Names: Fish Oil Concentrate; Natural Fish Oil
  Arms: Frozen capsule
Dietary Supplement: Capsule with food — Two room temperature fish oil capsules (300 mg EPA/DHA per capsule) by mouth three times daily with 8 ounces of water with food but no dairy products
  Other Names: Fish Oil Concentrate; Natural Fish Oil
  Arms: Capsule with food
Dietary Supplement: Capsule without food — Two room temperature fish oil capsules (300 mg EPA/DHA per capsule) by mouth three times daily with 8 ounces of water with no food or dairy products
  Other Names: Fish Oil Concentrate; Natural Fish Oil
  Arms: Capsule without food
Dietary Supplement: Capsule with milk — Two room temperature fish oil capsules (300 mg EPA/DHA per capsule) by mouth three times daily with 8 ounces of milk with no food or additional dairy products
  Other Names: Fish Oil Concentrate; Natural Fish Oil
  Arms: Capsule with milk

SUMMARY:
Many patients complain of fishy breath, upset stomach, or heartburn when taking the recommended amount of fish oil. A common recommendation made by pharmacists is to freeze the fish oil capsules to help decrease adverse gastrointestinal effects. Compliance with over-the-counter (OTC) fish oil is a concern considering the high number of capsules taken daily. The hypothesis of this study is that taking fish oil with milk will help lead to better patient compliance with no difference in adverse effects versus other administration methods.

DETAILED DESCRIPTION:
Fish oil has many proposed health benefits such as lowering triglycerides, decreasing inflammation, and reducing risk factors for cardiovascular disease. In order to take the recommended daily dose for hypertriglyceridemia using an OTC fish oil supplement, the daily recommended dose is at least 2 grams (2 capsules) three times a day. The American Heart Association recommends 2-4 grams of omega-3 fatty acid a day to aid in triglyceride reduction. Fish oil is known to cause GI-related adverse effects. Although reported to help, freezing fish oil capsules is inconvenient requiring access to a freezer three times a day. Currently there is a lack of literature to specify the best administration technique or patient compliance data for OTC fish oil supplements. The purpose of this study is to determine an ideal method of taking fish oil. This study will include up to 60 patients that are between the ages of 18-65 years who would be considered generally healthy. Patients will be recruited via e-mails sent to faculty and students of the School of Pharmacy, via flyers in Walgreen's stores, and through word of mouth. The patients will be randomly assigned to one of four treatment groups. Each treatment group will be given 180 capsules and instructed to take two capsules three times a day for thirty days with either food, no food, milk, or frozen. At the end of thirty days, the patient will return the bottle with any remaining pills to the investigator and take a survey. The investigators will assess compliance via pill count.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-65 years of age
* Minimal medication usage and controlled chronic health conditions

Exclusion Criteria:

* Patients with significant renal, hepatic, autoimmune or gastrointestinal tract disease
* Patients with uncontrolled chronic health conditions (e.g., diabetes, high blood pressure, high cholesterol or hypothyroidism)
* Receiving prescription anti-coagulation, prescription anti-platelet, prescription anti-inflammatory drugs, biologics, chronic steroids, chemotherapy, or otherwise excessive medication regimens
* Pregnant/nursing women, <18 years of age, prisoners, or the mentally ill

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Adverse Effects | 4 weeks
  Subjective survey based patient reported adverse effects

SECONDARY OUTCOMES:
Compliance | 4 weeks
  Pill count will be performed to assess medication compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Riche, Pharm.D., Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi School of Pharmacy, Jackson, Mississippi, United States

REFERENCES:
- [Background] Oelrich B, Dewell A, Gardner CD. Effect of fish oil supplementation on serum triglycerides, LDL cholesterol and LDL subfractions in hypertriglyceridemic adults. Nutr Metab Cardiovasc Dis. 2013 Apr;23(4):350-7. doi: 10.1016/j.numecd.2011.06.003. Epub 2011 Sep 15. PMID 21924882
- [Background] Eslick GD, Howe PR, Smith C, Priest R, Bensoussan A. Benefits of fish oil supplementation in hyperlipidemia: a systematic review and meta-analysis. Int J Cardiol. 2009 Jul 24;136(1):4-16. doi: 10.1016/j.ijcard.2008.03.092. Epub 2008 Sep 6. PMID 18774613
- [Background] Kris-Etherton PM, Harris WS, Appel LJ; American Heart Association. Nutrition Committee. Fish consumption, fish oil, omega-3 fatty acids, and cardiovascular disease. Circulation. 2002 Nov 19;106(21):2747-57. doi: 10.1161/01.cir.0000038493.65177.94. No abstract available. PMID 12438303
- [Background] Dietary supplementation with n-3 polyunsaturated fatty acids and vitamin E after myocardial infarction: results of the GISSI-Prevenzione trial. Gruppo Italiano per lo Studio della Sopravvivenza nell'Infarto miocardico. Lancet. 1999 Aug 7;354(9177):447-55. PMID 10465168
- [Background] Miller M, Stone NJ, Ballantyne C, Bittner V, Criqui MH, Ginsberg HN, Goldberg AC, Howard WJ, Jacobson MS, Kris-Etherton PM, Lennie TA, Levi M, Mazzone T, Pennathur S; American Heart Association Clinical Lipidology, Thrombosis, and Prevention Committee of the Council on Nutrition, Physical Activity, and Metabolism; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular Nursing; Council on the Kidney in Cardiovascular Disease. Triglycerides and cardiovascular disease: a scientific statement from the American Heart Association. Circulation. 2011 May 24;123(20):2292-333. doi: 10.1161/CIR.0b013e3182160726. Epub 2011 Apr 18. No abstract available. PMID 21502576
- [Background] Zabel R, Ash S, King N, Bauer J. Adherence to fish oil intervention in patients with chronic kidney disease. J Ren Nutr. 2010 Sep;20(5):329-33. doi: 10.1053/j.jrn.2010.01.003. Epub 2010 Mar 19. PMID 20303787
- [Derived] Malinowski SS, Barber KE, Kishk OA, Mays AA, Jones SR, Turner AL, Riche DM. Effect of fish oil supplement administration method on tolerability and adherence: a randomized pilot clinical trial. Pilot Feasibility Stud. 2019 Jan 8;5:3. doi: 10.1186/s40814-018-0387-0. eCollection 2019. PMID 30637118